CLINICAL TRIAL: NCT01787916
Title: Cross-over, Double-blind, Unicentric, 52 Week Trial of Liraglutide in Type 1 Diabetes.
Brief Title: 52 Week Trial of Liraglutide in Type 1 Diabetes
Acronym: LIDO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013LIDO
Record Dates: First submitted 2013-02-04; First posted 2013-02-11 (Estimated); Results first posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2014-03

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; overweight; insulin; liraglutide
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Overweight; Insulin Resistance | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide (Experimental): Liraglutide, s.c., 1.8 mg, die, 24 weeks
  Interventions: Drug: Liraglutide
- Placebo (Placebo Comparator): Liraglutide placebo (visually identical to study drug) will be given s.c. 1.8 mg for 24 weeks
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Liraglutide — Liraglutide will be compared to placebo for 24 weeks in a cross-over design
  Other Names: Victoza
  Arms: Liraglutide
Drug: Placebos — placebo will be compared to liraglutide for 24 weeks in a cross-over design
  Arms: Placebo

SUMMARY:
To our knowledge, no trial has specifically studied the effect of liraglutide combined with a basal/bolus insulin regimen in type 1 diabetes in a cross-over, double-blind, unicentric model. Moreover, the potential impact of a glucagon-like peptide-1 agonist on measures of abdominal fat (assessed by CT scan), insulin sensitivity (assessed by the gold standard euglycemic-hyperinsulinemic clamp) and satiety sensations have not been evaluated in this population.

Hypothesis Overweight participants with type 1 diabetes on liraglutide/insulin treatment will present improved glucose control with decreased HbA1c, decreased fasting and mean weekly glucose concentrations and glycemic excursions as well as increased insulin sensitivity compared to participants on placebo/insulin treatment. Participants with liraglutide/insulin treatment will also present improved endothelial function, lower body weight, central adipose tissue assessed by CT scan and higher satiety sensations assessed by visual analogue scales.

DETAILED DESCRIPTION:
Participants will be submitted to this double-blind cross-over protocol of 52-week use of liraglutide/placebo.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes non smoker BMI superior or equal to 25 diabetes duration superior or equal to 5 years

Exclusion Criteria:

* diabetic complication HbA1c superior or equal to 8.5% cancer acute or chronic pancreatitis

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley John Weisnagel, MD, Principal Investigator — CHU de Québec; Martin D'Amours, MD, Principal Investigator — CHU de Québec
Locations (1):
- CHU de Québec, Québec, Canada

IPD SHARING:
Plan to Share IPD: No
individual data will not be available to other researchers

REFERENCES:
- [Derived] Dube MC, D'Amours M, Weisnagel SJ. Beyond glycaemic control: A cross-over, double-blinded, 24-week intervention with liraglutide in type 1 diabetes. Diabetes Obes Metab. 2018 Jan;20(1):178-184. doi: 10.1111/dom.13063. Epub 2017 Sep 6. PMID 28722271

RESULTS

PARTICIPANT FLOW:
Groups:
- Liraglutide First, Then Placebo: Liraglutide, s.c., 1.8 mg, die, 24 weeks
  First Intervention (24 weeks)", "Washout (4 weeks)", and "Second Intervention (24 weeks
- Placebo First, the Liraglutide: subjects were submitted to placebo and liraglutide in a randomly manner
Period: First Intervention (24 Weeks)
Arm/Group | Liraglutide First, Then Placebo | Placebo First, the Liraglutide
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Washout (4 Weeks)
Arm/Group | Liraglutide First, Then Placebo | Placebo First, the Liraglutide
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Second Intervention (24 Weeks)
Arm/Group | Liraglutide First, Then Placebo | Placebo First, the Liraglutide
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Patients beginning with liraglutide will be switched to Placebo and vice versa
Arm/Group | All Study Participants
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Region of Enrollment [Number; unit: participants]
  Canada | 15

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Changes in Glycemic Control by HbA1c.
Description: To investigate the effect of 24 weeks of treatment with liraglutide combined with a basal/bolus insulin regimen in overweight participants with type 1 diabetes on glycemic control as assessed by HbA1c.
Time Frame: Measure changes in HbA1c at 24 and 52 weeks from baseline
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Groups:
- Placebo: Placebo visually identical to study drug will be given
  Liraglutide: Liraglutide will be compared to placebo for 24 weeks in a cross-over design
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 15 | 15
percentage of HbA1c | 0.3 (0.1) | 0.2 (0.1)

2. Secondary Outcome: Assessment of Changes on Adipose Tissue
Description: To investigate the effect of 24 weeks of treatment with liraglutide combined with the basal/bolus insulin regimen insulin on adipose tissue
Time Frame: Measure changes in the composite at 24 and 52 weeks from baseline
Reporting Status: Not Posted, anticipated posting 2017-12

ADVERSE EVENTS:
Time Frame: 1 yr
Arm/Group | Liraglutide | Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 13/15 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=15) | Placebo (N=15)
nausea (Gastrointestinal disorders) | 13 (13) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other